CLINICAL TRIAL: NCT03946072
Title: Multi-center Comparative Effectiveness Randomized Trial to Assess a Transseptal Approach to Left Ventricular Ablation Compared to Retrograde to Prevent Cerebral Emboli & Neurocognitive Decline in Adults With Ventricular Tachycardia/Premature Ventricular Contractions
Brief Title: Transseptal vs Retrograde Aortic Ventricular Entry to Reduce Systemic Emboli
Acronym: TRAVERSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TRAVERSE
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Neurocognitive Dysfunction
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transseptal Group (Active Comparator): Transseptal Aortic Approach Catheter Ablation Procedure
  Interventions: Procedure: Transseptal Aortic Approach Catheter Ablation Procedure
- Retrograde Group (Active Comparator): Retrograde Aortic Approach Catheter Ablation Procedure
  Interventions: Procedure: Retrograde Aortic Approach Catheter Ablation Procedure

INTERVENTIONS:
Procedure: Transseptal Aortic Approach Catheter Ablation Procedure — The transseptal approach entails obtaining femoral venous access, and, guided by fluoroscopy and intra-cardiac ultrasound, starting with a transseptal needle or radio frequency (RF) device inside the dilator of a long sheath; pulling down until the fossa ovalis in the interatrial septum is engaged on both fluoroscopy and intracardiac echo imaging; once on the left side, the long sheath is advanced over the transseptal needle, the needle and dilator are removed, and the ablation catheter can then be advanced across the mitral valve into the left ventricle.
  Arms: Transseptal Group
Procedure: Retrograde Aortic Approach Catheter Ablation Procedure — The retrograde aortic approach entails obtaining femoral arterial access and leaving a sheath in the femoral artery. Under fluoroscopy, an ablation catheter is then advanced up the ascending aorta where the catheter tip is curved using an internal mechanism controlled on the handle of the catheter to form a large loop (to prevent the tip from traveling down a coronary artery and causing trauma such as a dissection); the curved loop is advanced around the aortic arch and down the ascending aorta. To cross the aortic valve with this loop, the catheter is typically torqued in various directions until it falls through the aortic valve and into the left ventricle.
  Arms: Retrograde Group

SUMMARY:
This study is a prospective, multicenter, randomized (1:1) controlled comparative effectiveness trial of a transseptal approach to left ventricular ablation compared to a retrograde aortic approach to prevent cerebral emboli and neurocognitive decline in adults with ventricular tachycardia (VT) and/or premature ventricular contractions (PVCs).

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized (1:1) controlled comparative effectiveness trial of a transseptal approach to left ventricular ablation compared to a retrograde aortic approach to prevent cerebral emboli and neurocognitive decline in adults with ventricular tachycardia (VT) and/or premature ventricular contractions (PVCs). Participants will be followed for 6 months post-study procedure. This study will be conducted at up to 12 clinical sites in the United States. A total of one-hundred and fifty (150) participants will be enrolled and randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age
2. Planned/scheduled endocardial ventricular tachycardia (VT) or premature ventricular contraction (PVC) catheter ablation procedure
3. For this patient, the current plan of the operator must be to pursue a catheter ablation target in the left ventricular endocardium that can be accessed by either a transseptal puncture or retrograde aortic approach
4. Life expectancy of at least 1 year
5. Willing and able to undergo pre- and post-ablation MRIs
6. Willing and able to return and comply with scheduled follow up visits (through the 6 month follow-up)
7. Willing and able to provide written informed consent

Exclusion Criteria:

1. Planned epicardial ablation that would include a coronary angiogram (during the index ventricular tachycardia (VT) or premature ventricular contraction (PVC) catheter ablation procedure)
2. Any contraindication to MRI (as defined by the institution performing the MRI)
3. Clinical contraindication to a retrograde aortic approach as determined by the treating physician, including:

   1. Severe aortic stenosis
   2. Mechanical aortic valve
4. Clinical contraindication to a transseptal puncture as determined by the treating physician, including:

   1. Severe Mitral valve stenosis
   2. Mechanical Mitral valve
   3. Atrial septal defect (ASD) or Patent foramen ovale (PFO) closure device that would preclude a transseptal puncture
   4. Mitraclip or Alfieri mitral valve repair that would preclude a transseptal puncture
5. Planned or known need to perform either a retrograde aortic approach or transseptal approach (such as to target another site during the same procedure)
6. Inability to speak, read, and write in the English language at a 6th grade level (required for the Neurocognitive Function Testing)
7. Current mental impairment or other diagnosis which precludes accurate assessment of neurocognitive function or which may not allow patient to understand the nature, significance and scope of the study
8. Inability to perform neurocognitive function testing after > 24 hours free of sedating medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
cerebral embolic lesion incidence | on day 1 post-ablation
  incidence of new cerebral embolic lesions measured by magnetic resonance imaging (MRI) post-ablation as compared to pre-ablation imaging studies
overall neurocognitive function, change | from baseline (pre-ablation) to 6 months post-ablation
  percent change in overall neurocognitive function score from baseline (pre-ablation). The neurocognitive function examination includes items from the Brain Health Assessment, a validated, multi-domain testing battery aims to detect cognitive impairment in older adults. The TRAVERSE Testing Battery will include the following tests: Favorites (Forms A and B), Match (Forms A and B), Favorites Delay (Forms A and B), Favorites Recognition (Forms A and B), Dot Counting (Forms A and B), Flanker, and Running Dots.

SECONDARY OUTCOMES:
new cerebral embolic lesions, number | on day 1 post-ablation
  number of new cerebral embolic lesions per person, measured by magnetic resonance imaging (MRI) post-ablation as compared to pre-ablation imaging studies
complications related to the ablation procedure, rate | post-ablation, through Month 6
  rate of complications related to the ablation procedure
symptoms specific to VT/PVC, change | from pre-ablation to post-ablation, through Month 6
  change in self-reported symptoms specific to VT/PVC
quality of life composite score, change | from baseline (pre-ablation) to 6 months post-ablation
  change in quality of life score (composite summary points) measured using the Short Form 12-item Survey (SF-12), a validated measure of health status.
physical activity (MET-min/week), change | from baseline (pre-ablation) to 6 months post-ablation
  change in total physical activity (MET-min/week) measured using the International Physical Activity Questionnaire (IPAQ) short format questionnaire, validated for physical activity-related energy expenditure.
recurrent arrhythmias, rate | at 6 months post-ablation
  rate of recurrent arrhythmias determined as part of routine clinical care, measured using ECG and continuous ECG monitoring, if data is available

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Marcus, MD, Principal Investigator — University of California, San Francisco
Locations (21):
- United States (20):
  - Banner - University Medical Center, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Diego, San Diego, California
  - San Francisco Veterans Affairs (SFVA) Health Care, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Kaiser Permanente - Colorado, Aurora, Colorado
  - University of Colorado, Denver, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Washington University in St. Louis, St Louis, Missouri
  - Atrium Health/Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcus GM, Tung R, Gerstenfeld EP, Hue TF, Lin F, Cheng J, Weiss JP, Tzou WS, Hsia H, Ehdaie A, Cooper DH, Bunch TJ, Arkles J, Nazer B, Lee A, Hadjis A, Nguyen DT, Chelu MG, Moss J, Hsu JC, Valderrabano M, Bhave PD, Beaser AD, Kanagasundram A, Wazni O, Bradfield J, Wall G, Chang K, Yang M, Montenegro G, Jarrott S, Kramer JH, Kim AS, Morris YM, Dillon WP. Left Ventricular Entry to Reduce Brain Lesions During Catheter Ablation: A Randomized Trial. Circulation. 2025 Apr 15;151(15):1051-1059. doi: 10.1161/CIRCULATIONAHA.124.071352. Epub 2025 Feb 24. PMID 39989365